CLINICAL TRIAL: NCT06504160
Title: Safety and Efficacy of Topical Bacteriotherapy for Atopic Dermatitis Using Staphylococcus Hominis A9
Brief Title: Targeted Investigation of Microbiome 2 Treat Atopic Dermatitis (TIME-2)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (ADRN) (Unknown); Rho Federal Systems Division, Inc. (Industry); PPD, Thermo Fisher Scientific Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ADRN-14
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema; ADRN; TIME-2; microbiome; Staphylococcus hominis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ShA9 Topical Gel (Experimental): From Baseline to Week 2, ShA9 topical gel and TCS will be applied twice daily to areas selected at baseline, as well as any new lesions that arise. Once an area is treated, it will continue to be treated, regardless of lesional status.
  Clobetasol ointment will be applied immediately before the ShA9 in non-sensitive areas (e.g., arms). When necessary, fluocinonide ointment is a permissible alternative during this initial co-treatment. Hydrocortisone ointment will be applied with the ShA9 in sensitive areas (e.g., face).
  After two weeks of co-treatment, participants will continue using ShA9 without TCS for 12 more weeks. Participants will continue to apply ShA9 to any areas that received treatment during the first two weeks of the trial. If new lesions arise, these areas will also be treated. Once an area is treated, it will continue to be treated until the Week 14 visit regardless of lesional status.
  Interventions: Drug: ShA9 Topical Gel; Drug: Hydrocortisone Ointment; Drug: Clobetasol Ointment; Drug: Fluocinonide Ointment
- Placebo (Vehicle) Topical Gel (Placebo Comparator): From Baseline to Week 2, placebo (vehicle) topical gel and TCS will be applied twice daily to areas selected at baseline, as well as any new lesions that arise. Once an area is treated, it will continue to be treated, regardless of lesional status.
  Clobetasol ointment will be applied immediately before the placebo (vehicle) in non-sensitive areas (e.g., arms). When necessary, fluocinonide ointment is a permissible alternative during this initial co-treatment. Hydrocortisone ointment will be applied with the placebo (vehicle) in sensitive areas (e.g., face).
  After two weeks of co-treatment, participants will continue using placebo (vehicle) without TCS for 12 more weeks. Participants will continue to apply placebo (vehicle) to any areas that received treatment during the first two weeks of the trial. If new lesions arise, these areas will also be treated. Once an area is treated, it will continue to be treated until the Week 14 visit regardless of lesional status.
  Interventions: Drug: Hydrocortisone Ointment; Drug: Clobetasol Ointment; Drug: Fluocinonide Ointment; Drug: Placebo (Vehicle) Topical Gel

INTERVENTIONS:
Drug: ShA9 Topical Gel — The ShA9 topical gel contains phosphate-buffered saline solution (PBS), Glycerol, and hydroxyethylcellulose containing lyophilized ShA9 bacteria. The ShA9 bacteria is derived from a healthy donor-derived (allogeneic) commensal Staph species. The gel is manufactured and packaged by University of California San Diego (UCSD). It is applied twice daily to all areas identified as actively lesional during the Baseline Visit, regardless of ongoing lesional status, until the Week 14 Visit. If new lesions arise during this time, these areas will also be treated, regardless of ongoing lesional status, until the Week 14 Visit.
  Arms: ShA9 Topical Gel
Drug: Hydrocortisone Ointment — All participants will apply hydrocortisone ointment 2.5% alongside the study product in sensitive body areas (e.g., face, neck, intertriginous regions) for the first two weeks of the trial. It is applied twice daily to all areas identified as actively lesional during the Baseline Visit, regardless of ongoing lesional status, until the Week 2 Visit. If new lesions arise during this time, these areas will also be treated, regardless of ongoing lesional status, until the Week 2 Visit.
Drug: Clobetasol Ointment — All participants will apply clobetasol ointment 0.05% alongside the study product in non-sensitive body areas (e.g., arms, legs, torso) for the first two weeks of the trial. It will be applied twice daily to lesional skin and selected sampling areas from Baseline to Week 2. It is applied twice daily to all areas identified as actively lesional during the Baseline Visit, regardless of ongoing lesional status, until the Week 2 Visit. If new lesions arise during this time, these areas will also be treated, regardless of ongoing lesional status, until the Week 2 Visit.
Drug: Fluocinonide Ointment — Participants with a past intolerance to clobetasol or who become too sensitive to clobetasol in the initial two-week cotreatment period will apply fluocinonide ointment 0.05% as an alternative. In these cases, fluocinonide ointment 0.05% will be applied alongside the study product in non-sensitive body areas (e.g., arms, legs, torso) for the first two weeks of the trial. It is applied twice daily to all areas identified as actively lesional during the Baseline Visit, regardless of ongoing lesional status, until the Week 2 Visit. If new lesions arise during this time, these areas will also be treated, regardless of ongoing lesional status, until the Week 2 Visit.
Drug: Placebo (Vehicle) Topical Gel — The placebo (vehicle) topical gel contains phosphate-buffered saline solution (PBS), Glycerol, and hydroxyethylcellulose. The gel is manufactured and packaged by University of California San Diego (UCSD). It is applied twice daily to all areas identified as actively lesional during the Baseline Visit, regardless of ongoing lesional status, until the Week 14 Visit. If new lesions arise during this time, these areas will also be treated, regardless of ongoing lesional status, until the Week 14 Visit.
  Arms: Placebo (Vehicle) Topical Gel

SUMMARY:
This is a Phase 1b, randomized, placebo/vehicle-controlled, double-blinded, multi-center trial. It is designed to assess the safety and efficacy of S. hominis A9 (ShA9) topical application as a treatment for atopic dermatitis (AD). The trial will enroll adults and adolescents with atopic dermatitis who are culture positive for S. aureus colonization.

The primary safety objective of this study is to compare the safety profile of ShA9 to placebo (vehicle) over 14 weeks of application, which includes an initial two-week period of co-treatment with topical corticosteroids (TCS). The primary efficacy objective of this study is to assess the ability of ShA9, compared to placebo (vehicle), to prolong the period of atopic dermatitis control over 12 weeks after conclusion of an initial two-week period of co-treatment with TCS.

DETAILED DESCRIPTION:
Protocol ADRN-14 TIME-2 is a Phase 1b, randomized, placebo/vehicle-controlled, double-blinded, multi-center trial designed to assess the safety and efficacy of ShA9 topical application as a treatment for AD. This study will aim to enroll up to 86 participants; participants must be 12 years of age or older, have AD, and test culture positive for S. aureus (SA+) on their lesional skin.

An individual participant's involvement in this study will take approximately 20 weeks to complete, including approximately 2 weeks of screening, 14 weeks of treatment, and 4 weeks of safety follow-up.

An initial screening visit will be conducted to evaluate eligibility, including by assessing skin swabs collected from each participant for S. aureus positivity. SA+ participants will then begin an approximately 14-day period of standardized skin care by using over-the-counter products (e.g., Dove soap, Cetaphil moisturizer) which will be distributed from the study clinic. This is done to establish an informative baseline and allow for washout of any prohibited medications.

Participants who continue to meet eligibility criteria will then be randomized 1:1 to use either ShA9 gel or placebo (vehicle) gel for treatment of AD. Following randomization, for two weeks, each participant will receive co-treatment using TCS together with their assigned study product (active or placebo). Participants will then continue using their assigned study product without TCS for 12 more weeks. Participants will be seen in clinic approximately every 4 weeks during this time for sample/data collection and safety monitoring. Participants may be seen in clinic for additional visits to address any skin exacerbations while enrolled.

Participation concludes with a 4-week safety follow-up period during which use of ShA9 or placebo (vehicle) gel is halted. Participants will return to using over-the-counter products that will be distributed from the study clinic as needed, continuing to avoid prohibited medications and will be monitored for skin exacerbations or other adverse events.

ELIGIBILITY:
Inclusion Criteria:

Each individual must meet all of the following criteria at Screening to be eligible for enrollment as a study participant:

1. Must be able to understand and provide informed consent.
2. Male or female participant 12 years of age or older.
3. Meet ADRN Standard Diagnostic Criteria for active AD.

   Each individual must meet all of the following criteria at Baseline to be eligible for enrollment as a study participant:
4. Have at least 7 cm2 of lesional skin within the upper extremities, lower extremities, and/or trunk. Lesions on the face, neck, palms, soles, and intertriginous areas do not count toward the required area, as samples may not be taken from these areas. The required area may be one contiguous area or may be comprised of multiple areas with a compliant total area.
5. Have at least 3% body surface area of AD involvement as indicated by derived total area of involvement score during SCORAD assessment.
6. Have an IGA score of two or greater.
7. Have obtained skin swab test results prior to randomization indicating the presence of one positive S. aureus colonized lesion within the upper extremities, lower extremities, and/or trunk.
8. Each potential participant who can become pregnant must meet either of the following criteria prior to randomization to be eligible for enrollment as a study participant.

   1. Willing to remain abstinent from intercourse that may result in a pregnancy.
   2. Willing to use an FDA-approved method of contraception for the duration of study participation. Acceptable methods include the following:

      * Permanent sterilization of partner
      * Long-acting reversible contraceptives (e.g., intrauterine devices or systems, implantable rods, contraceptive injections) when used as directed for at least 7 days prior to Baseline.
      * Short-acting hormonal contraceptives (e.g., oral contraceptive pills, patch, vaginal ring) when used as directed for at least 30 days prior to Baseline
      * Barrier methods (e.g., condoms; diaphragm, sponge, or cervical cap with spermicide)

Exclusion Criteria:

Individuals who meet any of the following criteria at Screening or Baseline are not eligible for enrollment as study participants:

1. Inability or unwillingness to give written informed consent or comply with study protocol.
2. Has self-reported as pregnant or lactating during the Screening or Baseline Visit, or is pregnant as indicated by a positive pregnancy test result obtained at the Screening or Baseline Visit.
3. Sensitivity to or difficulty tolerating Dove fragrance-free bar soap, Cetaphil® lotion, alcohol-based cleaners, clobetasol and fluocinonide ointments, triamcinolone ointment, hydrocortisone ointment, glycerol, hydroxyethylcellulose or soy products.
4. Known recalcitrance to topical steroids, including class 1 steroids, within 6 months of the Screening Visit.
5. History of serious life-threatening reaction to tape or adhesives.
6. Known allergy to all antibiotics to which S. hominis A9 is sensitive. These include ampicillin-sulbactam, cefazolin, cefoxitin, clindamycin, daptomycin, doxycycline, levofloxacin, linezolid, minocycline, moxifloxacin, mupirocin, nitrofurantoin, oxacillin, rifampin, trimethoprim-sulfamethoxazole, and vancomycin.
7. Has a major defect in the epidermal barrier such as open wounds or genodermatoses (e.g., Netherton's syndrome).
8. Is immunocompromised (e.g., Human Immunodeficiency Virus (HIV)/Acquired Immunodeficiency Syndrome (AIDS), Wiskott-Aldrich Syndrome) or has an immune system disorder (e.g., autoimmune disease).
9. Has current malignant disease (except non-melanoma skin cancer in an area not affected by treatment).
10. Has a history of psychiatric disease or history of alcohol or drug abuse that, in the opinion of the study investigator, would interfere with the ability to comply with the study protocol.
11. Ongoing participation in another investigational trial or use of investigational drugs within 8 weeks, or five half-lives (if known), whichever is longer, of the Screening Visit.
12. Treatment with non-steroid systemic immunosuppressant within 6 months of the Screening Visit.
13. Treatment with any biologic, including dupilumab, within 16 weeks of the Screening Visit.
14. Treatment with oral or injectable therapy for AD (excluding oral steroids) within five half-lives (if known) or 16 weeks before the Screening Visit, whichever is longer.
15. Treatment with allergen immunotherapy within 30 days of Screening Visit.
16. Has close contacts (e.g., spouse, children, or members in the same household) who have severe barrier defects or are immunocompromised.
17. May, in the opinion of the investigator, have difficulty tolerating the medication washout requirements for topical AD treatments, prescription moisturizers, antibiotics, oral steroid therapies, and phototherapy ahead of Baseline.
18. Past or current medical conditions or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

    Individuals who meet any of the following criteria at Baseline are not eligible for enrollment as study participants:
19. Have more than 30% body surface area of AD involvement, as indicated by the derived total area of involvement score during SCORAD assessment.
20. Active bacterial, viral, or fungal skin infections, except for onychomycosis and tinea pedis.
21. Any noticeable breaks or cracks in the skin on the target areas of investigational product application, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection.
22. Use of topical AD treatments - including steroids and calcineurin inhibitors - on the upper extremities, lower extremities, or trunk within seven days of the Baseline Visit.
23. Treatment with prescription moisturizers classified as medical device (e.g., Atopiclair®, MimyX®, Epiceram®, etc.) on the upper extremities, lower extremities, or trunk within seven days of the Baseline Visit.
24. Use of any oral or topical antibiotic within fourteen days of the Baseline Visit.
25. Use of systemic corticosteroid therapies for any indication within 28 days of the Baseline Visit.
26. Use of systemic corticosteroid therapies for treatment of an asthma exacerbation within 3 months of the Baseline Visit.
27. Require a dose greater than 880 mcg/day of fluticasone propionate or equivalent inhaled corticosteroid to maintain asthma control, at the time of the Baseline Visit.
28. Any phototherapy for skin disease (such as narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + UVA [PUVA]) or regular use (more than 2 visits per week) of a tanning bed within 28 days of the Baseline Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-10-04 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Time to the first Atopic Dermatitis (AD) flare. | Week 2 (exclusive) through Week 14 (inclusive)
  Time (in days) to the first Atopic Dermatitis (AD) flare, indicated by having an Investigator Global Assessment (IGA) score that is greater than or equal to 2 and greater than the IGA score determined at Week 2. The IGA score is used to describe the overall appearance of AD lesions on a scale of 0 (clear) to 4 (severe).
Serious and non-serious treatment-emergent adverse events (TEAEs) related or possibly related to study treatment. | Baseline through Week 14
  The number of serious and non-serious treatment-emergent adverse events (TEAEs) related or possibly related to study treatment. If a participant experiences the same TEAE on multiple occasions, the event will be counted once for each occurrence when reporting the number of TEAEs.

SECONDARY OUTCOMES:
Serious and non-serious TEAEs related or possibly related to study treatment. | Week 14 (exclusive) through Week 18
  The number of serious and non-serious TEAEs related or possibly related to study treatment. If a participant experiences the same TEAE on multiple occasions, the event will be counted once for each occurrence when reporting the number of TEAEs.
Antibiotic sensitivity of S. aureus and S. epidermidis on the skin. | Baseline, Week 14
  The proportion of the skin bacteria, S. aureus and S. epidermidis, which can be isolated from skin swabs, that are sensitive to each of the following antibiotics: penicillin G, tetracycline, and erythromycin at Week 14 (post-ShA9 treatment) adjusted for the proportion of bacteria sensitive to antibiotic at Baseline.
Change in total Eczema Area and Severity Index (EASI) score. | Baseline, Week 14
  The change in total Eczema Area and Severity Index (EASI) score, which measures physical signs of atopic dermatitis, including area of involvement and severity (range: 0-72). Severity components include erythema, papulation, excoriation, and lichenification (0=absent, 1=mild, 2=moderate, 3=severe) for each body region (head/neck, trunk, arms, legs). Area of involvement (%) is assessed for each body region. Area and severity of each body region is weighted based on size of region, and region scores are added for a total EASI score (≤7=mild, >7 and ≤21.1=moderate, >21.1=severe). Descriptive note regarding time frame: if a participant was rescued with TCS within 14 days prior to their Week 14 visit, then their total EASI score at this timepoint will not be considered. Instead, the most recent total EASI score before the use of rescue TCS will be carried forward to represent Week 14.
EASI 50 | Baseline, Week 14
  The proportion of participants who achieve 50% or more reduction in their total EASI score. Descriptive note regarding time frame: if a participant was rescued with TCS within 14 days prior to their Week 14 visit, then their total EASI score at this timepoint will not be considered. Instead, the most recent total EASI score before the use of rescue TCS will be carried forward to represent Week 14.
EASI 75 | Baseline, Week 14
  The proportion of participants who achieve 75% or more reduction in their total EASI score. Descriptive note regarding time frame: if a participant was rescued with TCS within 14 days prior to their Week 14 visit, then their total EASI score at this timepoint will not be considered. Instead, the most recent total EASI score before the use of rescue TCS will be carried forward to represent Week 14.
Change in IGA score | Baseline, Week 14
  The change in IGA score. The IGA score is used to describe the overall appearance of AD lesions on a scale of 0 (clear) to 4 (severe). Descriptive note regarding time frame: if a participant was rescued with TCS within 14 days prior to their Week 14 visit, then their IGA score at this timepoint will not be considered. Instead, the most recent IGA score before the use of rescue TCS will be carried forward to represent Week 14.
Change in Pruritus Numeric Rating Scale (NRS) score. | Baseline, Week 14
  The change in Pruritus Numeric Rating Scale (NRS) score, which measures the average intensity of a pruritus (itch) during a 24-hour recall period on a scale of 0 (none) to 10 (worst imaginable itch). Descriptive note regarding time frame: if a participant was rescued with TCS within 14 days prior to their Week 14 visit, then their NRS score at this timepoint will not be considered. Instead, the most recent NRS score before the use of rescue TCS will be carried forward to represent Week 14.
Change in SCORing Atopic Dermatitis (SCORAD) score. | Baseline, Week 14
  The change in SCORing Atopic Dermatitis (SCORAD) score, which ranges from 0 (no AD) to 103 (severe). SCORAD is a composite index comprising a) the amount/extent of body surface area affected, b) subjective symptom visual analog assessments of itch and sleep loss, each on a scale of 0 (none) to 10 (worst imaginable), and c) 6 disease intensity assessments: dryness, erythema, edema/papulation, excoriation, lichenification and oozing/crusting, each graded from 0 (none) to 3 (severe). Descriptive note regarding time frame: if a participant was rescued with TCS within 14 days prior to their Week 14 visit, then their SCORAD score at this timepoint will not be considered. Instead, the most recent SCORAD score before the use of rescue TCS will be carried forward to represent Week 14.
Duration of rescue topical corticosteroid (TCS) use. | Week 2 (exclusive) through Week 14 (inclusive)
  The total number of days that topical corticosteroid (TCS) was used as a rescue medication within the upper extremities, lower extremities, and trunk of the body region, overall and separated by the potency class of steroids. The decision to begin the rescue TCS regimen due to skin exacerbation is dependent on investigator assessment, self-reported participant need, and standard of care.
Time to the first reported use of rescue TCS. | Week 2 (exclusive) through Week 14 (inclusive)
  Time (in days) to the first reported use of rescue TCS. The decision to begin the rescue TCS regimen due to skin exacerbation is dependent on investigator assessment, self-reported participant need, and standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallo, MD, PhD, Study Chair — University of California, San Diego: Dermatology Clinical Trials Unit; Tissa Hata, MD, Study Chair — University of California, San Diego: Dermatology Clinical Trials Unit; Donald Leung, MD, PhD, Study Chair — National Jewish Health: Division of Pediatric Allergy and Clinical Immunology
Locations (8):
- United States (8):
  - University of California, San Diego: Dermatology Clinical Trials Unit, San Diego, California
  - National Jewish Health: Division of Pediatric Allergy and Clinical Immunology, Denver, Colorado
  - Northwestern University Feinberg School of Medicine: Department of Dermatology, Chicago, Illinois
  - New York University Langone Health: Department of Pediatric Allergy and Immunology, New York, New York
  - Icahn School of Medicine at Mount Sinai: Department of Pediatrics Allergy & Immunology, New York, New York
  - University of Rochester Medical Center: Department of Dermatology, Rochester, New York
  - Cincinnati Children's Hospital Medical Center: Asthma Center, Cincinnati, Ohio
  - University of Wisconsin School of Medicine and Public Health: Division of Pediatric Allergy, Immunology and Rheumatology, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Share data upon study completion in Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: Post database lock
Access Criteria: Open Access
URL: http://www.immport.org/home

REFERENCES:
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/